CLINICAL TRIAL: NCT03742700
Title: Acute Health Effects of Short-term Use of E-cigarettes on Pulmonary and Cardiovascular System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Mateusz Jankowski, Principal Investigator, Medical University of Silesia
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: KNW/0022/KB1/37/I/17
Record Dates: First submitted 2018-11-11; First posted 2018-11-15 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: E-cigarette
Keywords: e-cigarette; health effects; cigarette smoking; exhaled nitric oxide; pulmonary function tests
MeSH Terms: conditions — Vaping; Cigarette Smoking | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Intervention Model Description: This was a laboratory-based intervention study: pre-post-post
Masking Description: Subjects were divided into 4 groups (n=30 each) based on their self-declared smoking status: control (C), tobacco cigarette smokers (T-Smokers), exclusive e-cigarette users (E-Smokers) and dual users (T/E-Smokers).
Oversight: FDA-regulated Device: No

ARMS (4):
- T-smokers (Experimental): T-smokers were asked to smoke a cigarette of one of the popular brands (0.6mg nicotine per one cigarette) according to their everyday habits.
  Interventions: Behavioral: Cigarette smoking
- E-smokers (Experimental): E-smokers were instructed to use e-cigarettes (12 mg/ml nicotine) in accordance with everyday habits for 5 minutes.
  Interventions: Behavioral: E-cigarette use
- T/E-smokers (Experimental): T/E-smokers (dual users) were instructed to use e-cigarettes (12 mg/ml nicotine) in accordance with everyday habits for 5 minutes.
  Interventions: Behavioral: E-cigarette use
- Control subjects (Placebo Comparator): The control subjects were asked to simulate the use of e-cigarettes (a device without e-liquid where aerosol was not created or inhaled).
  Interventions: Behavioral: Simulation of the use of e-cigarette

INTERVENTIONS:
Behavioral: Cigarette smoking — T-smokers were asked to smoke a cigarette of one of the popular brands (0.6mg nicotine per one cigarette) according to their everyday habits.
  Arms: T-smokers
Behavioral: E-cigarette use — E-smokers and dual users were instructed to use e-cigarettes (12 mg/ml nicotine) in accordance with everyday habits for 5 minutes.
  Arms: E-smokers; T/E-smokers
Behavioral: Simulation of the use of e-cigarette — The control subjects were asked to simulate the use of e-cigarettes (a device without e-liquid where aerosol was not created or inhaled).
  Arms: Control subjects

SUMMARY:
The goal of our study was to assess acute, short term respiratory (airflow, FeNO, O2 saturation, exhaled air temperature) and cardiovascular (heart rate, blood pressure) responses to smoking an e-cigarette in exclusive e-smokers and dual users and to compare these effects with responses to smoking a tobacco-cigarette in exclusive tobacco smokers.

ELIGIBILITY:
Inclusion Criteria:

- smoking status (cigarette or e-cigarette smoking)

Exclusion Criteria:

* occurrence of any chronic diseases,
* history of lung conditions (eg.: asthma or bronchial hyperactivity in childhood),
* presence of any allergic diseases,
* medication intake within the last 2 weeks,
* acute illnesses or infections in the last 2 weeks,
* influenza vaccination in the last 2 weeks,
* or current pregnancy or lactation.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
O2 saturation | pre - post (1 minute after exposure) - post (30 minute after exposure)
  The O2 measurement was made in the sitting position using the PULSOX 2 electronic pulse meter. The result was recorded 15 seconds after the start of the measurement.
Concentration of nitric oxide (FeNO) | pre - post (1 minute after exposure) - post (30 minute after exposure)
  FeNO measurements were made using the standard procedure in the sitting position with a clip attached to the nose using a NIOX MINO device for measuring fractional exhaled nitric oxide (FeNO). Subjects were instructed to breathe as deeply as possible through the mouthpiece to achieve maximum lung filling and then to exhale 50ml/sec for 10s. The measured FeNO values were expressed in ppb (parts per billion).
exhaled carbon monoxide (CO) | pre - post (1 minute after exposure) - post (30 minute after exposure)
  During the measurement, requirements regarding the length and intensity of the exhalation were taken into account. The measurements were made using the PiCo Smokylyzer device. The measured CO levels were expressed in ppm (parts per million).
temperature of exhaled air | pre - post (1 minute after exposure) - post (30 minute after exposure)
  The measurement was made using the standard procedure in the sitting position using an X-Halo Breath Thermometer [20]. Respondents were instructed to breathe according to the procedure recommended by the device manufacturer. The temperature of exhaled air was expressed in Celsius degrees (°C).
spirometric testing | pre - post (1 minute after exposure) - post (30 minute after exposure)
  Airflow and lung volume were measured in the sitting position with a noseclip according to the ATS/ERS guidelines. The measurements were made using the EasyOne 2001 spirometer and included FEV1, FVC, FEV1% FVC, PEF and MEF75,50,25. Expiratory maneuvers were repeated until a minimum of three technically correct, repeatable measurements were obtained.
heart rate | pre - post (1 minute after exposure) - post (30 minute after exposure)
  Heart rate was measured in the sitting position, the result of measurement was expressed in beats per minute.
blood pressure | pre - post (1 minute after exposure) - post (30 minute after exposure)
  Blood pressure was measured in the sitting position, the result of measurement was expressed in mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Grzegorz Brożek, MD, PhD, Study Director — Department of Epidemiology, School of Medicine in Katowice, Medical University of Silesia in Katowice, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: E-smoking: Emerging public health problem? — http://ijomeh.eu/E-smoking-Emerging-public-health-problem-,67520,0,2.html